



# The Effects of Preoperative Blood Flow Restriction Training in Patients Undergoing ACL Reconstruction

# **RESEARCH PACKAGE**

| Patient Contact: • Email: |
|----------------------------|
| • Email: |
| • Cell: |

## **Protocol Version 2.0:**

October 28, 2022

## **Principle Investigator:**

Resident Physician, Division of Orthopaedic Surgery, University of Toronto

## **Primary Supervisor:**

Staff Orthopaedic Surgeon, Mount Sinai Hospital, Toronto, ON

# Table of Contents

- 1. Consent Form
- 2. Patient Demographics
- 3. Methods / BFR Study Design
- 4. Training Load Conversion Chart
- 5. Participation Checklist
- 6. Pre Intervention KOOS Questionnaire
- 7. Post Intervention KOOS Questionnaire
- 8. Pre Intervention SF-12 Questionnaire
- 9. Post Intervention SF-12 Questionnaire



#### CONSENT TO PARTICIPATE IN A RESEARCH STUDY

**Study Title:** The Effects of Preoperative Blood Flow Restriction Training in Patients Undergoing ACL Reconstruction

INVESTIGATORS:

Study Coordinator: Division of Orthopaedics, Department of Surgery,

Women's College Hospital, Toronto, Ontario

(416) 323-7526

#### Introduction

You are being asked to take part in a research study. Please read this explanation about the study and its risks and benefits before you decide if you would like to take part. You should take as much time as you need to make your decision. You should ask the study doctor or study staff to explain anything that you do not understand and make sure that all of your questions have been answered before signing this consent form. Before you make your decision, feel free to talk about this study with anyone you wish. Participation in this study is voluntary.

## **Background and Purpose**

You are being asked to consider participating in this research study because you have a tear of your anterior cruciate ligament, and are electing to undergo anterior cruciate ligament reconstruction (ACLR) surgery. The purpose of the study is to explore the potential effect that pre-surgery physiotherapy with blood flow restriction training may have on improving the strength and function of your injured knee/leg.

## **Background:**

The anterior cruciate ligament (ACL) is one of the most important ligaments in the knee as it controls joint stability. It is also one of the most commonly injured ligaments in young adults. ACL injury can result in joint instability and restriction of activities, even with physiotheraphy and other conservative treatment. Anterior cruciate ligament reconstruction (ACLR) is the surgical repair of this torn ligament, and can be done using 3 different grafts from the patients own body; the patellar tendon, the hamstring tendon, and the quadriceps tendon. All 3 graft types are commonly used, and your surgeon will have chosen the graft type they believed was best for you after examining you in clinic.

The quadricep femoris (QF) is a large group of muscle in the front of your thigh, muscle strength plays an important role in rehabilitation and overall outcome after lower limb injury or surgery. Weakening of this muscle group is common in patients with anterior cruciate ligament (ACL) injuries undergoing ACL reconstruction due to prior inactivity before surgery. In order to combat the challenges of the weakening of the quads muscle for patients with an ACL injury,

physiotherapy and in particular blood flow restriction (BFR) training during physiotherapy has been shown to have potential benefits for patients after their surgery. This method of treatment can help reduce the amount of quadriceps weakening by allowing muscles to maintain their strength and size while performing low load exercises. This is important as it is normally very difficult to rehabilitate these muscles with a painful and injured knee. Our study would like investigate, whether or not this form of training is beneficial prior to surgery so that patient's enter their operation with improved strength and function setting themselves up for success in the post operative period. If this study is able to demonstrate a positive outcome for patients prior to their surgery, blood flow restriction will prove to be a valuable training modality for all patients awaiting ACL reconstruction.

## Study Design

If you consent to participate in this study, you will still receive normal standard of care treatment for your injury, no care will be denied. Your involvement in this study will last from the date you consent to participate during your appointment with your treating doctor to book surgery, until the week of your surgery. This time frame will vary depending on how far away the date of your surgery is, however the actual active time spent doing activities for this study will only be the 4 weeks leading up to your day of surgery.

In taking part in this study, you will be asked to participate in 4 weeks of physiotherapy, with 3 x 30 minute sessions per week for a total of 12 sessions, this will occur in the 4 weeks leading up to your surgery day. This is a randomized study, meaning participants will be randomized to one of two study groups for investigation. You will have a 50/50 chance of being randomized to either group, like the flip of a coin. Group 1, the experimental group, will have participants complete the course of pre-operative physiotherapy sessions while using blood flow restriction cuffs during their physiotherapy exercises, while group 2, the non-experimental group, will complete the same physiotherapy sessions but will not be using any additional devices during the exercises. All other study activities remain the same regardless of which group you have been randomized to.

You will also be asked to undergo physical examination of your knee including range of motion and strength testing, performed both manually by your care team, and on a machine called a Biodex. You will also be asked to complete two questionnaires that ask about the daily functioning ability of your knee, and your general health. These questionnaires and physical tests will only be done twice, once on the first day of your physiotherapy, and again on the last day of your physiotherapy. There are no study activities that take place after your surgery.

These physiotherapy sessions and strength testing sessions will be provided to you at no cost, however you may experience costs related to time and transit to attend these sessions. Every effort will be made to book these sessions on dates and times most convenient to you and your schedule.

The study team will consult your medical records to collect information such as your medical history and demographics (e.g., gender, date of birth) and take notes of the relevant information (data) for this research study.

## Risks Related to Being in the Study

This study does not change any of the risks of treatment(s) that you may receive as part of your care. Blood flow restriction has been extensively reviewed and poses no greater risk than traditional heavy-low training. All patients will be appropriately screened for

general health conditions that may impact their ability to participate in the project (e.g heart conditions, diabetes or severe high blood pressure). This study involves physical exercises and exams that if done correctly do not pose any significant risk, and will be supervised by medical professionals.

## Benefits to Being in the Study

While you should not expect any direct benefits from participating in this study, it is possible benefits may exist from undergoing pre-operative physiotherapy. The data you provide during this study may have an impact on future outcomes for ACL reconstruction and this could help future patients who have an ACL tear.

## **Voluntary Participation**

Your participation in this study is voluntary. You may decide not to be in this study, or to be in the study now and then change your mind later. You may leave the study at any time without affecting your care You may refuse to answer any question you do not want to answer, or not answer an interview question by saying "pass".

We will give you new information that is learned during the study that might affect your decision to stay in the study.

#### Alternatives to Being in the Study

You do not have to participate in this study to continue to receive treatment for your anterior cruciate ligament tear. Full standard care will be provided to you regardless of your involvement in this study.

## Confidentiality

If you agree to join this study, the study doctor and his/her study team will look at your personal health information and collect only the information they need for the study. Personal health information is any information that could be used to identify you and includes your:

- name.
- address,
- date of birth,
- new or existing medical records, that includes types, dates and results of medical tests or procedures.

The information that is collected for the study will be kept in a locked and secure area by the study doctor for 7 years. Only the study team or the people or groups listed below will be allowed to look at your records. Your participation in this study also may be recorded in your medical record at this hospital.

The following people may come to the hospital to look at the study records and at your personal health information to check that the information collected for the study is correct and to make sure the study followed proper laws and guidelines:

- Representatives of the study organizing committee.
- Mount Sinai Hospital Research Ethics Board.

All information collected during this study, including your personal health information, will be kept confidential and will not be shared with anyone outside the study unless required by law. Any information about you that is sent out of the hospital will have a code and will not show your name or address, or any information that directly identifies you. You will not be named in any reports, publications, or presentations that may come from this study.

If you decide to leave the study, the information about you that was collected before you left the study will still be used. No new information will be collected without your permission.

## In Case You Are Harmed in the Study

If you become ill, injured or harmed as a result of taking part in this study, you will receive care. The reasonable costs of such care will be covered for any injury, illness or harm that is directly a result of being in this study. In no way does signing this consent form waive your legal rights nor does it relieve the investigators, sponsors or involved institutions from their legal and professional responsibilities. You do not give up any of your legal rights by signing this consent form.

## **Expenses Associated with Participating in the Study**

You will not have to pay for any of the procedures involved with this study. You will not be reimbursed for transportation, meals, time, inconvenience, etc.

#### **Conflict of Interest**

The investigators have an interest in completing this study. Their interests should not influence your decision to participate in this study. You should not feel pressured to join this study.

## **Communication with Your Family Doctor**

Your family doctor may be informed that you are taking part in this study so that your study doctor and family doctor can help you make informed decisions about your medical care.

## **Questions About the Study**

If you have any questions, concerns or would like to speak to the study team for any reason, please call: Dr. John Theodoropoulos at 416 586 4800, Ext. 8699 or the Study Coordinator, Shgufta Docter at 416-323-6400, Ext 7526

If you have any questions about your rights as a research participant or have concerns about this study, call Ronald Heslegrave, Ph. D., Chair of the Mount Sinai Hospital Research Ethics Board (REB) or the Research Ethics office number at 416-586-4875. The REB is a group of people who oversee the ethical conduct of research studies. These people are not part of the study team. Everything that you discuss will be kept confidential.

## Consent

| This study has been explained to me I know that I may leave the study at a the use of my personal health inform | any time. I agree to take | part in this study {and to |
|---|---|---|
| Print Study Participant's Name | Signature | <br>Date |
| (You will be given a signed copy of the | nis consent form) | |
| My signature means that I have explanate answered all questions | ained the study to the pa | articipant named above. I |
| Print Name of Person Obtaining Con | sent Signature | <br>Date |
| Was the participant assisted during t | he consent process? | YES NO |
| If YES, please check the relevant bo | x and complete the sign | ature space below: |
| ☐ The person signing below acted a process and attests that the study as has had any questions answered. | • | . • |
| Print Name of Translator | Signature | <br>Date |
| Relationship to Participant | Language | |
| ☐ The consent form was read to the the study as set out in this form was questions answered. | | |
| Print Name of Witness | Signature | Date |
| Relationship to Participant | | |

| Patient Demographics | | |
|----------------------------------------------|---------------------|-------|
| NAME: | | |
| AGE: | | |
| GENDER (circle): MALE | FEMALE | OTHER |
| WEIGHT (lbs): | | |
| LEG DOMINANCE: RIGHT | LEFT | |
| E.g. If you were to kick a soccer ball, whic | h foot would you ch | oose? |
| OCCUPATION: | | |
| PRIMARY SPORT: | | |
| PAST MEDICAL CONDITIONS: | | _ |
| MEDICATIONS: | | |

## Methods/Study Design

## **Group Allocation**:

- Patients will be randomized into 1 of 2 groups:
  - o **BFR Group**: BFR Physiotherapy Pre Operatively (16 patients)
  - o **Non-BFR Group:** Same Physiotherapy protocol without BFR intervention Pre Operatively (16 patients)
- This will be a balanced randomization using an online randomization tool.

#### **Inclusion Criteria**:

- Sagittal Knee instability caused by ACL tear requiring surgical reconstruction
- Minimum 4 weeks since the time of injury
- Age 18 to 50 years
  - o Range of motion required
    - Active extension deficit <5°, Active flexion > 120°
  - No previous surgery to affected knee

#### **Exclusion Criteria:**

- Functional impairment (neuro disease, gait abnormality, ambulatory aids at baseline)
- Severe spine or lower limb injuries
- Comorbidities including cardiovascular, respiratory or metabolic disease, blood coagulation disorders, current smoker

#### **BFR Cuff Details:**

- 14 cm wide contoured pneumatic tourniquet cuff (Delfi Easi-Fit Contour Thigh Cuff)
- Estimate best tourniquet fit based on patient's thigh circumference
  - RED = 18"
  - GREEN = 24'
  - BLUE = 34"
- Placed around proximal thigh, connected to portable pressure regulating system (Delfi Portable Tourniquet System)
- Inflated to 80% LOP (Limb Occlusion Pressure) automatically performed with Delfi System

## BFR Exercise Protocol: To be completed at Mt. Sinai Hospital

- Patient will perform a total of 12 sessions prior to surgery (3 sessions/week x 4 weeks)
- Patients will perform single leg knee extension exercise in a closed kinetic chain on a leg-press machine.
- Non injured leg will not perform any exercises but will act as control and be measured for strength and clinical outcome
- Patients in the non BFR group will perform the same protocol but there will be no inflation of their tourniquet during testing
- Load will be individually set to 15% 1RM for warm up and 25% 1RM for intervention
  - O Warmup: 10 to 15 reps at 15% 1RM workload, no BFR occlusion
    - Rest: 30 seconds
  - o 1st Set: cuff inflated to 80% LOP, patient completes 30 reps at 25% 1 RM
    - Rest: 30 seconds
  - o 2<sup>nd</sup> Set: cuff remains inflated to 80% LOP, patient completes 15 reps at 25% 1RM
    - Rest: 30 seconds
  - o 3<sup>rd</sup> Set: cuff remains inflated to 80% LOP, patient completes 15 reps at 25% 1RM
    - Rest: 30 seconds
    - 4<sup>th</sup> Set: cuff remains inflated to 80% LOP, patient completes 15 reps at 25% 1RM
      - Session complete, cuff deflated.
- Load Progression
  - o If patient's are able to complete all 75 repetitions (30-15-15-15) on two consecutive sessions, their load will be increased by 10% at the subsequent session

# **Training Load Conversion Chart**

| TRAINING LOAD CHART | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Max reps (RM) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 |
| % 1RM | 100% | 95% | 93% | 90% | 87% | 85% | 83% | 80% | 77% | 75% | 70% |
| Load | 10 | 9.5 | 9.3 | 9 | 8.7 | 8.5 | 8.3 | 8 | 7.7 | 7.5 | 7 |
| | 20 | 19 | 18.6 | 18 | 17.4 | 17 | 16.6 | 16 | 15.4 | 15 | 14 |
| | 30 | 28.5 | 27.9 | 27 | 26.1 | 25.5 | 24.9 | 24 | 23.1 | 22.5 | 21 |
| | 40 | 38 | 37.2 | 36 | 34.8 | 34 | 33.2 | 32 | 30.8 | 30 | 28 |
| | 50 | 47.5 | 46.5 | 45 | 43.5 | 42.5 | 41.5 | 40 | 38.5 | 37.5 | 35 |
| | 60 | 57 | 55.8 | 54 | 52.2 | 51 | 49.8 | 48 | 46.2 | 45 | 42 |
| | 70 | 66.5 | 65.1 | 63 | 60.9 | 59.5 | 58.1 | 56 | 53.9 | 52.5 | 49 |
| | 80 | 76 | 74.4 | 72 | 69.6 | 68 | 66.4 | 64 | 61.6 | 60 | 56 |
| | 90 | 85.5 | 83.7 | 81 | 78.3 | 76.5 | 74.7 | 72 | 69.3 | 67.5 | 63 |
| | 100 | 95 | 93 | 90 | 87 | 85 | 83 | 80 | 77 | 75 | 70 |
| | 110 | 104.5 | 102.3 | 99 | 95.7 | 93.5 | 91.3 | 88 | 84.7 | 82.5 | 77 |
| | 120 | 114 | 111.6 | 108 | 104.4 | 102 | 99.6 | 96 | 92.4 | 90 | 84 |
| | 130 | 123.5 | 120.9 | 117 | 113.1 | 110.5 | 107.9 | 104 | 100.1 | 97.5 | 91 |
| | 140 | 133 | 130.2 | 126 | 121.8 | 119 | 116.2 | 112 | 107.8 | 105 | 98 |
| | 150 | 142.5 | 139.5 | 135 | 130.5 | 127.5 | 124.5 | 120 | 115.5 | 112.5 | 105 |
| | 160 | 152 | 148.8 | 144 | 139.2 | 136 | 132.8 | 128 | 123.2 | 120 | 112 |
| | 170 | 161.5 | 158.1 | 153 | 147.9 | 144.5 | 141.1 | 136 | 130.9 | 127.5 | 119 |
| | 180 | 171 | 167.4 | 162 | 156.6 | 153 | 149.4 | 144 | 138.6 | 135 | 126 |
| | 190 | 180.5 | 176.7 | 171 | 165.3 | 161.5 | 157.7 | 152 | 146.3 | 142.5 | 133 |
| | 200 | 190 | 186 | 180 | 174 | 170 | 166 | 160 | 154 | 150 | 140 |
| | 210 | 199.5 | 195.3 | 189 | 182.7 | 178.5 | 174.3 | 168 | 161.7 | 157.5 | 147 |
| | 220 | 209 | 204.6 | 198 | 191.4 | 187 | 182.6 | 176 | 169.4 | 165 | 154 |
| | 230 | 218.5 | 213.9 | 207 | 200.1 | 195.5 | 190.9 | 184 | 177.1 | 172.5 | 161 |
| | 240 | 228 | 223.2 | 216 | 208.8 | 204 | 199.2 | 192 | 184.8 | 180 | 168 |
| | 250 | 237.5 | 232.5 | 225 | 217.5 | 212.5 | 207.5 | 200 | 192.5 | 187.5 | 175 |
| | 260 | 247 | 241.8 | 234 | 226.2 | 221 | 215.8 | 208 | 200.2 | 195 | 182 |
| | 270 | 256.5 | 251.1 | 243 | 234.9 | 229.5 | 224.1 | 216 | 207.9 | 202.5 | 189 |
| | 280 | 266 | 260.4 | 252 | 243.6 | 238 | 232.4 | 224 | 215.6 | 210 | 196 |
| | 290 | 275.5 | 269.7 | 261 | 252.3 | 246.5 | 240.7 | 232 | 223.3 | 217.5 | 203 |
| | 300 | 285 | 279 | 270 | 261 | 255 | 249 | 240 | 231 | 225 | 210 |
| | 310 | 294.5 | 288.3 | 279 | 269.7 | 263.5 | 257.3 | 248 | 238.7 | 232.5 | 217 |
| | 320 | 304 | 297.6 | 288 | 278.4 | 272 | 265.6 | 256 | 246.4 | 240 | 224 |
| | 330 | 313.5 | 306.9 | 297 | 287.1 | 280.5 | 273.9 | 264 | 254.1 | 247.5 | 231 |
| | 340 | 323 | 316.2 | 306 | 295.8 | 289 | 282.2 | 272 | 261.8 | 255 | 238 |
| | 350 | 332.5 | 325.5 | 315 | 304.5 | 297.5 | 290.5 | 280 | 269.5 | 262.5 | 245 |
| | 360 | 342 | 334.8 | 324 | 313.2 | 306 | 298.8 | 288 | 277.2 | 270 | 252 |
| | 370 | 351.5 | 344.1 | 333 | 321.9 | 314.5 | 307.1 | 296 | 284.9 | 277.5 | 259 |
| | 380 | 361 | 353.4 | 342 | 330.6 | 323 | 315.4 | 304 | 292.6 | 285 | 266 |
| | 390 | 370.5 | 362.7 | 351 | 339.3 | 331.5 | 323.7 | 312 | 300.3 | 292.5 | 273 |
| | 400 | 380 | 372 | 360 | 348 | 340 | 332 | 320 | 308 | 300 | 280 |
| | 410 | 389.5 | 381.3 | 369 | 356.7 | 348.5 | 340.3 | 328 | 315.7 | 307.5 | 287 |
| | 420 | 399 | 390.6 | 378 | 365.4 | 357 | 348.6 | 336 | 323.4 | 315 | 294 |
| | 430 | 408.5 | 399.9 | 387 | 374.1 | 365.5 | 356.9 | 344 | 331.1 | 322.5 | 301 |
| | 440 | 418 | 409.2 | 396 | 382.8 | 374 | 365.2 | 352 | 338.8 | 330 | 308 |
| | 450 | 427.5 | 418.5 | 405 | 391.5 | 382.5 | 373.5 | 360 | 346.5 | 337.5 | 315 |
| | 460 | 437 | 427.8 | 414 | 400.2 | 391 | 381.8 | 368 | 354.2 | 345 | 322 |
| | 470 | 446.5 | 437.1 | 423 | 408.9 | 399.5 | 390.1 | 376 | 361.9 | 352.5 | 329 |
| | 480 | 456 | 446.4 | 432 | 417.6 | 408 | 398.4 | 384 | 369.6 | 360 | 336 |
| | 490 | 465.5 | 455.7 | 441 | 426.3 | 416.5 | 406.7 | 392 | 377.3 | 367.5 | 343 |
| | 500 | 475 | 465 | 450 | 435 | 425 | 415 | 400 | 385 | 375 | 350 |

- Training load chart can be used to calculate estimated 1-repetion maximum (1RM) values from multiple repetitions completed
  - For example, if an athlete completes 8 repetitions of the squat at 160 lbs, the estimated 1RM would be 200 lbs.
- Training load chart can also be used to assign intensity percentages for program design
  - For examaple, if an athlete's 1RM for the squat is 200 lbs, he/she should be able to successfully complete 10 repetitions of 150 lbs, or 75% max intensity.

# **Participation Checklist**

| | Date | Supervisor | Completed | Comments |
|---|---|---|---|---|
| Patient Randomization | | Lawrence Wengle | Y/N | BFR Group or CONTROL Group |
| Pre Intervention Biodex | | Paul Papoutsakis | Y/N | |
| Pre Intervention Scores | | | Y/N | KOOS and SF-12 Questionnaires |
| BFR Session 1 | | | Y / N | 10RM = 1RM = Thigh circumferencemm |
| BFR Session 2 | | | Y / N | |
| BFR Session 3 | | | Y / N | |
| BFR Session 4 | | | Y / N | |
| BFR Session 5 | | | Y / N | |
| BFR Session 6 | | | Y/N | |
| BFR Session 7 | | | Y/N | |
| BFR Session 8 | | | Y / N | |
| BFR Session 9 | | | Y/N | |
| BFR Session 10 | | | Y / N | |
| BFR Session 11 | | | Y / N | |
| BFR Session 12 | | | Y / N | Thigh circumferencemm |
| Post Intervention Biodex | | Paul Papoutsakis | Y/N | |
| Post Intervention Scores | | | Y / N | KOOS and SF-12 Questionnaires |
| ACL Surgery | | Dr. Theodoropoulos | Y/N | |

| | KOOS | S KNEE S | URVEY | | |
|---|---|---|---|---|---|
| Today's date: | | Date of b | oirth:/ | / | |
| Name: | | | | | |
| information will<br>well you are ab<br>Answer every o | help us keep t<br>le to perform yo<br>question by tick<br>u are unsure ab | rack of how you<br>ur usual activitie<br>ing the appropr | ມ feel about yo<br>s.<br>iate box, only | t your knee. The<br>our knee and ho<br>one box for eac<br>n, please give th | ow<br>ch |
| Symptoms These question the last week. | ns should be an | swered thinking | of your knee | symptoms durii | าg |
| S1. Do you have<br>Never | swelling in your larely | knee? Sometimes | Often | Always | |
| S2. Do you feel g<br>moves?<br>Never | grinding, hear clic<br>Rarely | Sometimes | often | nen your knee Always | |
| S3. Does your kr<br>Never | nee catch or hang Rarely | up when moving? Sometimes | Often | Always | |
| S4. Can you strai<br>Always | ighten your knee i<br>Often | fully? Sometimes | Rarely | Never | |
| S5. Can you bend<br>Always | d your knee fully?<br>Often | Sometimes | Rarely | Never | |
| experienced du | uring the last v | | nee. Stiffness | iffness you havis is a sensation knee joint. | |
| S6. How severe i | is your knee joint Mild | stiffness after firs<br>Moderate | t wakening in th<br>Severe | e morning? Extreme | |
| S7. How severe in None | is your knee stiffn<br>Mild | ness after sitting, ly<br>Moderate | ying or resting la<br>Severe | ater in the day? Extreme | |

| <b>Pain</b><br>P1. How often do<br><sup>Never</sup> □ | you experience Monthly | e knee pain?<br>Weekly | Daily | Always | |
|---|---|---|---|---|---|
| What amount of | | have you experie | enced the last | week during th | е |
| P2. Twisting/pivo | oting on your kr<br>Mild | nee<br>Moderate | Severe | Extreme | |
| P3. Straightening None | knee fully<br>Mild | Moderate | Severe | Extreme | |
| P4. Bending knee None | fully<br>Mild | Moderate | Severe | Extreme | |
| P5. Walking on fl<br>None | at surface Mild | Moderate | Severe | Extreme | |
| P6. Going up or d<br>None | lown stairs<br>Mild | Moderate | Severe | Extreme | |
| P7. At night while<br>None | e in bed<br>Mild | Moderate | Severe | Extreme | |
| P8. Sitting or lyin None | g<br>Mild | Moderate | Severe | Extreme | |
| P9. Standing upri<br>None | ght<br>Mild | Moderate | Severe | Extreme | |
| ability to move | uestions conc<br>around and<br>indicate the | ern your physical<br>to look after you<br>degree of difficu | ırself. For eac | h of the followin | ıg |
| A1. Descending s None | tairs<br>Mild | Moderate | Severe | Extreme | |
| A2. Ascending sta | airs<br>Mild | Moderate | Severe | Extreme | |

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| A3. Rising from None | om sitting<br>Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| A4. Standing None | Mild | Moderate | Severe | Extreme |
| A5. Bending None | to floor/pick up an o<br>Mild | object<br>Moderate | Severe | Extreme |
| A6. Walking None | on flat surface<br>Mild | Moderate | Severe | Extreme |
| A7. Getting in None | n/out of car<br>Mild | Moderate | Severe | Extreme |
| A8. Going sh<br>None | opping<br>Mild<br><b>□</b> | Moderate | Severe | Extreme |
| A9. Putting o | n socks/stockings<br>Mild | Moderate | Severe | Extreme |
| A10. Rising f | From bed Mild | Moderate | Severe | Extreme |
| A11. Taking None | off socks/stockings Mild | Moderate | Severe | Extreme |
| A12. Lying in<br>None | n bed (turning over,<br>Mild | maintaining knee Moderate | position) Severe | Extreme |
| A13. Getting None | in/out of bath<br>Mild<br>□ | Moderate | Severe | Extreme |
| A14. Sitting None | Mild<br>□ | Moderate | Severe | Extreme |
| A15. Getting None | on/off toilet Mild | Moderate | Severe | Extreme |

a of

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| A16. Heavy domestic duties (moving heavy boxes, scrubbing floors, etc) | | | | | |
|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | Extreme |
| ۸17 | Light domostic | dutica (cooking | ducting ata) | | |
| | Light domestic ( | Mild | Moderate | Severe | Extreme |
| • | | | | D | |
| | _ | _ | _ | _ | _ |
| The f | er level. The o | ions concern<br>questions sho | nal activities<br>your physical fur<br>ould be answered<br>uring the last we | d thinking of w | hat degree |
| | | • | J | • | |
| | Squatting<br>None | Mild | Moderate | Severe | Extreme |
| | _ | _ | _ | _ | _ |
| SP2. | Running | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| SP3. | Jumping | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| an | | | | | |
| | Twisting/pivotin | | | C | F . |
| - | None | Mild<br>□ | Moderate | Severe | Extreme |
| | ш | ш | Ц | Ц | ш |
| SP5 | Kneeling | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| • | | | | | |
| Qual | ity of Life | | | | |
| | - | u avvera of vou | r knoo problem? | | |
| | | Monthly | r knee problem?<br>Weekly | Daily | Constantly |
| | _ | _ | _ | _ | _ |
| Q2. Have you modified your life style to avoid potentially damaging activities to your knee? | | | | | |
| No | ot at all | Mildly | Moderately | Severely | Totally |
| | | | h lack of confidenc | | |
| No | ot at all | Mildly | Moderately | Severely | Extremely |
| 04.1 | | | da | | |
| _ | n general, how n<br>None | Mild | do you have with y Moderate | your knee?<br>Severe | Extreme |
| - | | | Moderate | Severe | |

Thank you very much for completing all the questions in this questionnaire.

| KOOS KNEE SURVEY | | | | | |
|---|---|---|---|---|---|
| Today's date: | | Date of b | oirth:/ | / | |
| Name: | | | | | |
| information will<br>well you are ab<br>Answer every o | help us keep t<br>le to perform yo<br>question by tick<br>u are unsure ab | rack of how you<br>ur usual activitie<br>ing the appropr | ມ feel about yo<br>s.<br>iate box, only | t your knee. The<br>our knee and ho<br>one box for eac<br>n, please give th | ow<br>ch |
| Symptoms These question the last week. | ns should be an | swered thinking | of your knee | symptoms durii | าg |
| S1. Do you have<br>Never | swelling in your larely | knee? Sometimes | Often | Always | |
| S2. Do you feel g<br>moves?<br>Never | grinding, hear clic<br>Rarely | Sometimes | often | nen your knee Always | |
| S3. Does your kr<br>Never | nee catch or hang Rarely | up when moving? Sometimes | Often | Always | |
| S4. Can you strai<br>Always | ighten your knee i<br>Often | fully? Sometimes | Rarely | Never | |
| S5. Can you bend<br>Always | d your knee fully?<br>Often | Sometimes | Rarely | Never | |
| experienced du | uring the last v | | nee. Stiffness | iffness you havis is a sensation knee joint. | |
| S6. How severe i | is your knee joint Mild | stiffness after firs<br>Moderate | t wakening in th<br>Severe | e morning? Extreme | |
| S7. How severe in None | is your knee stiffn<br>Mild | ness after sitting, ly<br>Moderate | ying or resting la<br>Severe | ater in the day? Extreme | |

| <b>Pain</b><br>P1. How often do<br><sup>Never</sup> □ | you experience Monthly | e knee pain?<br>Weekly | Daily | Always | |
|---|---|---|---|---|---|
| What amount of | | have you experie | enced the last | week during th | е |
| P2. Twisting/pivo | oting on your kr<br>Mild | nee<br>Moderate | Severe | Extreme | |
| P3. Straightening None | knee fully<br>Mild | Moderate | Severe | Extreme | |
| P4. Bending knee None | fully<br>Mild | Moderate | Severe | Extreme | |
| P5. Walking on fl<br>None | at surface<br>Mild | Moderate | Severe | Extreme | |
| P6. Going up or d<br>None | lown stairs<br>Mild | Moderate | Severe | Extreme | |
| P7. At night while<br>None | e in bed<br>Mild | Moderate | Severe | Extreme | |
| P8. Sitting or lyin None | g<br>Mild | Moderate | Severe | Extreme | |
| P9. Standing upri<br>None | ght<br>Mild | Moderate | Severe | Extreme | |
| ability to move | uestions conc<br>around and<br>indicate the | ern your physical<br>to look after you<br>degree of difficu | ırself. For eac | h of the followin | g |
| A1. Descending s None | tairs<br>Mild | Moderate | Severe | Extreme | |
| A2. Ascending sta | airs<br>Mild | Moderate | Severe | Extreme | |

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| A3. Rising from None | om sitting<br>Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| A4. Standing None | Mild | Moderate | Severe | Extreme |
| A5. Bending None | to floor/pick up an o<br>Mild | object<br>Moderate | Severe | Extreme |
| A6. Walking None | on flat surface<br>Mild | Moderate | Severe | Extreme |
| A7. Getting in None | n/out of car<br>Mild | Moderate | Severe | Extreme |
| A8. Going sh<br>None | opping<br>Mild<br><b>□</b> | Moderate | Severe | Extreme |
| A9. Putting o | n socks/stockings<br>Mild | Moderate | Severe | Extreme |
| A10. Rising f | From bed Mild | Moderate | Severe | Extreme |
| A11. Taking None | off socks/stockings Mild | Moderate | Severe | Extreme |
| A12. Lying in<br>None | n bed (turning over,<br>Mild | maintaining knee Moderate | position) Severe | Extreme |
| A13. Getting None | in/out of bath<br>Mild<br>□ | Moderate | Severe | Extreme |
| A14. Sitting None | Mild<br>□ | Moderate | Severe | Extreme |
| A15. Getting None | on/off toilet Mild | Moderate | Severe | Extreme |

a of

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| A16. Heavy domestic duties (moving heavy boxes, scrubbing floors, etc) | | | | | |
|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | Extreme |
| ۸17 | Light domostic | dutica (cooking | ducting ata) | | |
| | Light domestic ( | Mild | Moderate | Severe | Extreme |
| • | | | | D | |
| | _ | _ | _ | _ | _ |
| The f | er level. The o | ions concern<br>questions sho | nal activities<br>your physical fur<br>ould be answered<br>uring the last we | d thinking of w | hat degree |
| | | • | J | • | |
| | Squatting<br>None | Mild | Moderate | Severe | Extreme |
| | _ | _ | _ | _ | _ |
| SP2. | Running | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| SP3. | Jumping | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| an | | | | | |
| | Twisting/pivotin | | | C | F . |
| - | None | Mild<br>□ | Moderate | Severe | Extreme |
| | ш | ш | Ц | Ц | ш |
| SP5 | Kneeling | | | | |
| | None | Mild | Moderate | Severe | Extreme |
| • | | | | | |
| Qual | ity of Life | | | | |
| | - | u avvera of vou | r knoo problem? | | |
| | | Monthly | r knee problem?<br>Weekly | Daily | Constantly |
| | _ | _ | _ | _ | _ |
| Q2. Have you modified your life style to avoid potentially damaging activities to your knee? | | | | | |
| No | ot at all | Mildly | Moderately | Severely | Totally |
| | | | h lack of confidenc | | |
| No | ot at all | Mildly | Moderately | Severely | Extremely |
| 04.1 | | | da | | |
| _ | n general, how n<br>None | Mild | do you have with y Moderate | your knee?<br>Severe | Extreme |
| - | | | Moderate | Severe | |

Thank you very much for completing all the questions in this questionnaire.

# SF-12 Health Survey

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. **Answer each question by choosing just one answer**. If you are unsure how to answer a question, please give the best answer you can.

| 1. In general, would you say you | health is: | | | | | |
|---|---|---|---|---|---|---|
| □₁ Excellent □₂ Very good | □₃ Good | □₄ Fair | | □₅ Poor | | |
| The following questions are about | | | ng a typica | | your health now | <del></del> |
| <u>limit you</u> in these activities? If so | | g.ii. uo uu | | uuy. 2000 | your mount more | = |
| | | YES, | | VEC | NO not | |
| | | limited<br>a lot | | YES,<br>limited<br>a little | NO, not<br>limited<br>at all | |
| <ol><li>Moderate activities such as moving<br/>a vacuum cleaner, bowling, or p</li></ol> | | □1 | | □2 | □3 | |
| 3. Climbing <b>several</b> flights of stairs | i. | □1 | | <b>□</b> 2 | Пз | |
| During the <u>past 4 weeks,</u> have yo<br>daily activities <u>as a result of your</u> | | | oblems wit | th your work | or other regula | r |
| | | | YES | | NO | |
| <ol> <li>Accomplished less than you w</li> </ol> | vould like. | | □1 | | □2 | |
| 5. Were limited in the <b>kind</b> of work | or other activities | S. | □1 | | □2 | |
| During the <u>past 4 weeks,</u> have yo<br>daily activities <u>as a result of any</u> | | | | | | r |
| | | | YES | | NO | |
| 6. Accomplished less than you w | ould like. | | □1 | | <b>□</b> 2 | |
| 7. Did work or activities less caref | ully than usual. | | □1 | | □2 | |
| B. During the <u>past 4 weeks</u> , how he home and housework)? | much <u>did pain ir</u> | <u>nterfere</u> with | our norm | al work (incl | uding work outs | ide |
| □₁ Not at all □₂ A little bit | □₃ Mode | erately | □₄ Quite | a bit | □₅ Extremely | |
| These questions are about how y<br>For each question, please give the<br>How much of the time during the | ne one answer th | | | | ve been feeling. | |
| | All of<br>the<br>time | Most<br>of the<br>time | A good<br>bit of<br>the time | Some of the time | A little<br>of the<br>time | Non<br>of th<br>time |
| 9. Have you felt calm & peaceful? | □1 | □2 | □3 | □4 | □5 | □6 |
| 0. Did you have a lot of energy? | □1 | □2 | Пз | □4 | □5 | □6 |
| Have you felt down-hearted and blue? | □1 | □2 | Пз | □4 | □5 | □6 |
| 12. During the <u>past 4 weeks</u> , how interfered with your social activit | | | | | onal problems | |

# SF-12 Health Survey

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. **Answer each question by choosing just one answer**. If you are unsure how to answer a question, please give the best answer you can.

| 1. In general, w | ould you say your l | nealth is: | | | | | |
|---|---|---|---|---|---|---|---|
| □₁ Excellent | □₂ Very good | □₃ Good | □₄ Fair | | □₅ Poor | | |
| | uestions are about se activities? If so, | | might do duri | ng a typic | al day. Does <u>y</u> | our health now | |
| <u>you</u> o. | | | | | | | |
| | | | YES,<br>limited<br>a lot | | YES,<br>limited<br>a little | NO, not<br>limited<br>at all | |
| | vities such as moving<br>eaner, bowling, or pla | | □1 | | <b>□</b> 2 | □3 | |
| 3. Climbing sev | reral flights of stairs. | | □1 | | <b>□</b> 2 | Пз | |
| | <u>t 4 weeks,</u> have you<br>as a result of your <sub>l</sub> | | | oblems wi | th your work o | or other regular | <u> </u> |
| | | | | YES | | NO | |
| - | ned less than you wo | | | □1 | | □2 | |
| | in the <b>kind</b> of work | | | □1 | | □2 | |
| | <u>t 4 weeks,</u> have you<br>as a result of any e | | | | | | |
| | | | | YES | | NO | |
| | ed less than you wo | | | □1 | | □2 | |
| | ctivities less careful | • | | □1 | | □2 | |
| 8. During the p<br>the home and h | <u>ast 4 weeks</u> , how n<br>nousework)? | iuch <u>did pain i</u> | nterfere with y | our norm | al work (inclu | ding work outsi | de |
| □₁ Not at all | □₂ A little bit | □₃ Mod | erately | □₄ Quite | a bit | □₅ Extremely | |
| | ns are about how yo<br>ion, please give the | | | | | e been feeling. | |
| How much of th | ne time during the $\underline{r}$ | ast 4 weeks | | | | | |
| | | All of<br>the<br>time | Most of the time | A good<br>bit of<br>the time | Some of the time | A little of the time | None of the time |
| 9. Have you felt o | alm & peaceful? | □1 | □2 | Пз | □4 | □5 | □6 |
| 10. Did you have a | a lot of energy? | □1 | □2 | Пз | □4 | □5 | □6 |
| 11. Have you felt of blue? | down-hearted and | □1 | □2 | Пз | □4 | □5 | □6 |
| | <u>past 4 weeks,</u> how r<br>your social activitie | | | | | nal problems | |
| □₁ All of the time | All of the time $\Box_2$ Most of the time $\Box_3$ Some of the time $\Box_4$ A little of the time $\Box_5$ None of the time | | | | | | |